CLINICAL TRIAL: NCT03289455
Title: A Single-Arm, Open-Label, Multi-Centre, Phase I/II Study Evaluating the Safety and Clinical Activity Of AUTO3, a CAR T Cell Treatment Targeting CD19 And CD22 in Paediatric And Young Adult Patients With Relapsed or Refractory B Cell Acute Lymphoblastic Leukaemia
Brief Title: CD19 /22 CAR T Cells (AUTO3) for the Treatment of B Cell Acute Lymphoblastic Leukemia (ALL)
Acronym: AMELIA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTO3-PA1; 2016-004680-39 (EudraCT Number)
Record Dates: First submitted 2017-09-11; First posted 2017-09-21 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: B Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Refractory Childhood Acute Lymphoblastic Leukemia; B-cell Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukaemia; CD19 Positive; CD22 Positive; Relapsed Acute Lymphoblastic Leukaemia; Refractory Acute Lymphoblastic Leukaemia; AUTO3
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AUTO3 (Experimental): Paediatric patients with relapse or refractory B-cell ALL
  Interventions: Biological: AUTO3 (CD19/22 CAR T cells

INTERVENTIONS:
Biological: AUTO3 (CD19/22 CAR T cells — Following preconditioning with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with 1 to 5.0 x 10⁶/kg CD19/CD22 Chimeric Antigen Receptor (CAR) positive T cells as a single or split dose.

SUMMARY:
The purpose of this study is to test the safety and efficacy of AUTO3, a CAR T cell treatment targeting CD19 and CD22 in paediatric or young adult patients with relapsed or refractory B cell acute lymphoblastic leukaemia.

DETAILED DESCRIPTION:
The study will consist of 2 phases, a Phase I or dose escalation phase and a Phase II or expansion phase. Paediatric or young adult patients with relapsed or refractory B cell ALL will be enrolled in both phases of the study. Eligible patients will undergo leukapheresis in order to harvest T cells, which is the starting material for the manufacture of the autologous CAR T product AUTO3 which is a CD19 and CD22 dual targeting CAR T cell product. Following pre-conditioning by a chemotherapeutic regimen, the patient will receive AUTO3 intravenously as a single or split dose and will then enter a 24-month follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female patients aged 1-24 years with high risk (HR) relapsed/refractory B-lineage ALL, AND:

   1. Any bone marrow (BM) relapse or central nervous system (CNS) relapse with detectable BM disease after allogeneic stem cell transplant (SCT) and must be ≥6 months from SCT at the time of AUTO3 infusion; OR,
   2. HR first relapse; OR,
   3. Standard risk relapse patients with HR cytogenetics; OR,
   4. Second or greater relapse; OR,
   5. BM minimal residual disease (MRD) ≥10-³ prior to planned SCT; OR,
   6. Any on-treatment relapse in patients aged 16-24 years.

      (Phase II Only - Criteria in addition to those described above:)
   7. Primary refractory disease; OR,
   8. Patients with Philadelphia chromosome positive ALL are eligible if they are intolerant to or have failed 2 lines of tyrosine kinase inhibitor (TKI) therapy, or if TKI therapy is contraindicated; OR,
   9. Isolated CNS relapse but with ≤CNS Grade 2 disease at time of enrolment.
2. Documentation of CD19 and or CD22 expression on leukaemic blasts in the BM, peripheral blood, or cerebrospinal fluid within 3 months of screening.
3. Detectable disease in the BM at a level ≥10-⁴ (Phase I only).
4. Absolute lymphocyte count ≥0.5 x 10⁹/L.
5. Adequate renal, hepatic, pulmonary, and cardiac function.
6. Karnofsky (age ≥10 years) or Lansky (age <10 years) score ≥50%.
7. Willing and able to give written, informed consent to the current study (patient and/or parent or legal guardian).

Exclusion Criteria:

1. Isolated extra-medullary disease relapse.
2. Active CNS involvement of ALL (CNS Grade 3 per National Comprehensive Cancer Network guidelines).
3. Active infectious bacterial or viral disease requiring IV anti-microbials for treatment.
4. Females who are pregnant or lactating.
5. Females of child-bearing potential and post pubertal male participants who are unwilling to use highly effective methods of contraception for a period of 1 year after the AUTO3 infusion.
6. Inability to tolerate leukapheresis.
7. Prior CD19 or CD22 targeted therapy with Grade 4 toxicity or ≥refractory Grade 3 cytokine release syndrome (CRS) or ≥Grade 3 drug related CNS toxicity.
8. Pre-existing significant neurological disorder.
9. Stem Cell Transplant patients only: active significant acute graft versus host disease (GVHD) or moderate/severe chronic GVHD requiring systemic steroids or other immunosuppressant within 4 weeks of enrolment.
10. The following medications are excluded:

    1. Steroids: Therapeutic doses of steroids must be stopped >72 hours prior to AUTO3 infusion and leukapheresis. However, physiological replacement doses of steroids are allowed: <12 mg/m2/day hydrocortisone or equivalent.
    2. Allogeneic cellular therapy: Any donor lymphocyte infusions must be completed >6 weeks prior to AUTO3 infusion.
    3. Graft versus host disease therapies: Any drug used for GVHD must be stopped >4 weeks prior to AUTO3 infusion.
    4. Chemotherapy: Should be stopped 1 week prior to leukapheresis and 2 days prior to starting pre-conditioning chemotherapy.
11. Known allergy to albumin, dimethyl sulfoxide, cyclophosphamide or fludarabine.

For AUTO3 Infusion: Patients meeting any of the following exclusion criteria will not be treated with AUTO3 or treatment will be delayed until they no longer meet these criteria:

1. Severe intercurrent infection.
2. Requirement for supplementary oxygen.
3. Allogeneic transplant recipients with active significant acute GVHD overall Grade ≥II or moderate/severe chronic GVHD requiring systemic steroids.

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Royal Manchester Children's Hospital, Manchester

REFERENCES:
- [Derived] Roddie C, Lekakis LJ, Marzolini MAV, Ramakrishnan A, Zhang Y, Hu Y, Peddareddigari VGR, Khokhar N, Chen R, Basilico S, Raymond M, Vargas FA, Duffy K, Brugger W, O'Reilly MA, Wood L, Linch DC, Peggs KS, Bachier C, Budde EL, Lee Batlevi C, Bartlett N, Irvine D, Tholouli E, Osborne W, Ardeshna KM, Pule MA. Dual targeting of CD19 and CD22 with bicistronic CAR-T cells in patients with relapsed/refractory large B-cell lymphoma. Blood. 2023 May 18;141(20):2470-2482. doi: 10.1182/blood.2022018598. PMID 36821767

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 patients were screened, 20 patients leukapheresed and 15 patients were pre-conditioned with cyclophosphamide and fludarabine and infused with AUTO3 at 3 different dose levels.
Groups:
- 1x10^6 CD19/CD22 CAR-positive T Cells/kg: Patients assigned in this Cohort received actual doses of 0.3 to 2x10^6 CD19/CD22 CAR-positive T cells
- 3x10^6 CD19/CD22 CAR-positive T Cells/kg: All patients assigned in this Cohort received actual doses of 3x10^6 CD19/CD22 CAR-positive T cells
- 5x10^6 CD19/CD22 CAR-positive T Cells/kg: Patients assigned in this Cohort received actual doses of 4.3 to 5x10^6 CD19/CD22 CAR-positive T cells
Period: Overall Study
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Started | 4 | 5 | 6
Completed | 0 (Completed = Received AUTO3 infusion and completed 24 months visit) | 0 (Completed = Received AUTO3 infusion and completed 24 months visit) | 0 (Completed = Received AUTO3 infusion and completed 24 months visit)
Not Completed | 4 | 5 | 6
Not completed — Death | 1 | 0 | 0
Not completed — Sponsor decision due to covid19 restrictions | 0 | 1 | 0
Not completed — No CART persistence in MRD negativity. Patient proceeded with HSCT | 0 | 0 | 1
Not completed — Progressive disease | 3 | 4 | 5

BASELINE CHARACTERISTICS:
Population: Patients infused with AUTO3
Groups:
- Total: Total of all reporting groups
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg | Total
Number analyzed (Participants) | 4 | 5 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 6 | 15
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 4
  Male | 4 | 3 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 5 | 6 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 5 | 6 | 15
Karnofsky/Lansky score [Median (Full Range); unit: percentage] — The Karnofsky and Lansky scales are used to determine changes in daily activities for patients aged 10 to 24 years and <10 years, respectively. The Karnofsky scale ranges from 0% (death) to 100% (normal, co complaints, no signs of disease) and the Lansky scale from 0% (unresponsive) to 100% (fully active, normal).
  percentage | 95 [80 to 100] | 90 [80 to 100] | 100 [90 to 100] | 90 [80 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grade 3-5 Toxicities Occurring Within the Dose Limiting Toxicity (DLT) Period of AUTO3 Infusion
Time Frame: Within 30 days (+/- 3 days) after the last dose of AUTO3.
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set)
Measure: Count of Participants; unit: Participants
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 4 | 5 | 6
Participants | 4 | 4 | 6

2. Primary Outcome: Number of Patients With Dose Limiting Toxicity (DLT) of AUTO3
Description: DLT was defined as i) any new non-hematological adverse event (AE) of Grade 3 or higher toxicity using the NCI CTCAE (version 5.0), which was probably or definitely related to AUTO3 therapy, which occurred within the DLT evaluation period, and which failed to resolve to Grade 2 or better within 14 days, despite appropriate supportive measures; ii) Grade 4 cytokine release syndrome (CRS) or neurotoxicity, cerebral edema, or Grade 3 neurotoxicity (including cerebral edema) that lasted >72 hours; iii) Grade >3 disseminated intravascular coagulation; iv) Grade >2 infusion reaction; v) Any other fatal event (Grade 5) or life-threatening event (Grade 4) that could not be managed with conventional supportive measures or which in the opinion of the Safety Evaluation Committee (SEC) necessitated dose reduction or other modification to trial treatment to avoid a similar hazard in future patients.
Time Frame: Within 30 days (+/- 3 days) after the last dose of AUTO3.
Measure: Count of Participants; unit: Participants
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 4 | 5 | 6
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Patients Achieving Morphological Remission (Complete Response(CR) or Complete Response With Incomplete Count Recovery (CRi) and Minimal Residual Disease (MRD)-Negative Response in the Bone Marrow (PCR)).
Description: Morphological response evaluations were based on the response criteria for ALL according to the NCCN guidelines version 2.2014. Minimal residual disease-negative status was achieved if MRD was <10^-4 (0.01%) by PCR amplification of individual rearrangements of Ig genes and/or flow cytometry MRD testing.
Time Frame: Within 30 days (+/- 3 days) post AUTO3 infusion
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set).
Measure: Count of Participants; unit: Participants
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 4 | 5 | 6
Participants | 3 | 5 | 5

4. Secondary Outcome: Feasibility of Generating AUTO3: Number of Patients' Cells Successfully Manufactured as a Proportion of the Number of Patients Undergoing Leukapheresis
Description: Feasibility of product generation was examined by assessing the number of AUTO3 successfully manufactured as a fraction of the number of patients undergoing leukapheresis (all patients screened).
Time Frame: Up to 8 weeks post leukapheresis
Population: Patients who underwent leukapheresis. This outcome is measured before patients received infusion with AUTO3. Therefore, no split by dose cohort can be provided.
Measure: Count of Participants; unit: Participants
Groups:
- AUTO3: Pediatric and young adult patients with relapsed or refractory B cell ALL
Arm/Group | AUTO3
Number analyzed (Participants) | 20
Participants | 19

5. Secondary Outcome: Event-Free Survival (EFS) by Morphological Analysis
Description: Time from date of first AUTO3 infusion until the earliest of treatment failure (defined as not achieving CR/CRi post AUTO3 infusion / no response), morphological relapse, or death due to any cause, whichever occurred first.
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 4 | 5 | 6
months | 3.48 [0.03 to NA] — Upper limit of the confidence interval was not reached | 12.42 [3.94 to NA] — Upper limit of the confidence interval was not reached | 2.79 [0.03 to NA] — Upper limit of the confidence interval was not reached

6. Secondary Outcome: Number of Patients With CD19- and/or CD22-negative Relapse
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial dose) of AUTO3 and had morphological relapses
Measure: Count of Participants; unit: Participants
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 2 | 3 | 4
Participants | 0 | 2 | 1

7. Secondary Outcome: Relapse-Free Survival (RFS) by Morphological Analysis
Description: Time from first achievement of morphological CR/CRi post AUTO3 treatment until the earliest of morphological relapse, or death due to any cause, whichever occurred first.
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 4 | 5 | 6
months | 6.09 [2.56 to NA] — Upper limit of the confidence interval was not reached | 11.50 [3.02 to NA] — Upper limit of the confidence interval was not reached | 3.98 [1.87 to NA] — Upper limit of the confidence interval was not reached

8. Secondary Outcome: Overall Survival (OS)
Description: Calculated from the date of AUTO3 treatment to the date of death anytime post AUTO3 infusion. Patients who had not died were censored at the date of last contact.
Time Frame: Up to 2 years after the last patient was infused
Population: Patients who received at least 1 (complete or partial) dose of AUTO3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 4 | 5 | 6
months | 10.17 [2.30 to NA] — The upper limit of the confidence interval was not reached | 25.20 [4.34 to NA] — The upper limit of the confidence interval was not reached | NA [4.07 to NA] — The median was not estimable. The upper limit of the confidence interval was not reached

9. Secondary Outcome: Expansion of AUTO3 Following Adoptive Transfer
Description: Expansion of AUTO3 was measured as the median peak (Cmax) of transgene levels in the peripheral blood after AUTO3 infusion
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 and had evaluable cellular kinetics data (who had at least 1 cellular kinetics concentration post AUTO3 infusion above the lower limit of quantitation) (cellular kinetics analysis set)
Measure: Median (Full Range); unit: vector copies/ug DNA
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 4 | 5 | 4
vector copies/ug DNA | 10240 [5690 to 37000] | 102000 [34800 to 127000] | 79800 [13200 to 104000]

10. Secondary Outcome: Persistence of AUTO3 Following Adoptive Transfer
Description: Persistence of AUTO3 was measured by quantitative polymerase chain reaction (qPCR) and/or flow cytometry at a range of time points in the peripheral blood and the bone marrow.
  Persistence was defined as the timepoint in days of last detectable CAR T cell by qPCR or last assessment if zero copies per μg DNA (whichever occurred later) before morphological relapse (Tlast).
Time Frame: Up to 2 years
Population: as for outcome 9
Measure: Median (Full Range); unit: days
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 4 | 5 | 4
days | 41.7 [19.8 to 256.8] | 343.7 [62.7 to 538.9] | 24.3 [18.8 to 570.8]

11. Secondary Outcome: Duration of B Cell Aplasia
Description: Depletion of circulating B cells assessed by flow cytometry at a range of time points in the peripheral blood
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of the pre-conditioning regimen (safety set)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
Number analyzed (Participants) | 4 | 5 | 6
months | NA [NA to NA] — B cell aplasia from the database was inconclusive because the total lymphocytes from the peripheral blood analyzed by flow cytometry were not collected systematically | NA [NA to NA] — B cell aplasia from the database was inconclusive because the total lymphocytes from the peripheral blood analyzed by flow cytometry were not collected systematically | NA [NA to NA] — B cell aplasia from the database was inconclusive because the total lymphocytes from the peripheral blood analyzed by flow cytometry were not collected systematically

ADVERSE EVENTS:
Time Frame: From AUTO3 infusion (Day 0) until the end of study (2 years after last patient dosed) or withdrawal, whichever occurred first
Arm/Group | 1x10^6 CD19/CD22 CAR-positive T Cells/kg | 3x10^6 CD19/CD22 CAR-positive T Cells/kg | 5x10^6 CD19/CD22 CAR-positive T Cells/kg
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/5 | 3/6
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/5 | 3/6
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1x10^6 CD19/CD22 CAR-positive T Cells/kg (N=4) | 3x10^6 CD19/CD22 CAR-positive T Cells/kg (N=5) | 5x10^6 CD19/CD22 CAR-positive T Cells/kg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1x10^6 CD19/CD22 CAR-positive T Cells/kg (N=4) | 3x10^6 CD19/CD22 CAR-positive T Cells/kg (N=5) | 5x10^6 CD19/CD22 CAR-positive T Cells/kg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (4) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (6) | 3 (9) | 5 (16)
Catheter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingival abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parvovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Human herpes virus 6 serology positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (4)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (24) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (6)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early completion of the study leading to small numbers of patients analyzed from the Phase I part of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT03289455/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT03289455/SAP_001.pdf